CLINICAL TRIAL: NCT02143648
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel, 3-Arm Study of the Safety and Anti-Pruritic Efficacy of Nalbuphine HCl ER Tablets in Hemodialysis Patients With Uremic Pruritus
Brief Title: Study of Nalbuphine HCl ER Tablets in Hemodialysis Patients With Uremic Pruritus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR02; 2013-005625-22 (EudraCT Number)
Record Dates: First submitted 2014-05-17; First posted 2014-05-21 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Uremic Pruritus; Pruritus
Keywords: uremic; pruritus; itch; chronic itch; nalbuphine
MeSH Terms: conditions — Pruritus | interventions — BID protein, human; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- nalbuphine HCl ER 60mg (Experimental): nalbuphine HCl ER tablets 60 mg BID
  Interventions: Drug: nalbuphine HCl ER tablets 60 mg BID
- nalbuphine HCl ER 120mg (Experimental): nalbuphine HCl ER tablets 120 mg BID
  Interventions: Drug: nalbuphine HCl ER tablets 120mg BID
- Sugar pill (Placebo Comparator): Placebo tablets BID
  Interventions: Drug: Placebo tablets BID

INTERVENTIONS:
Drug: nalbuphine HCl ER tablets 60 mg BID — nalbuphine HCl ER tablets 60 mg BID administered for 6 weeks
  Other Names: nalbuphine ER
  Arms: nalbuphine HCl ER 60mg
Drug: nalbuphine HCl ER tablets 120mg BID — nalbuphine HCl ER tablets 120mg BID administered for 6 weeks
  Other Names: nalbuphine ER
  Arms: nalbuphine HCl ER 120mg
Drug: Placebo tablets BID — Placebo tablets BID administered for 8 weeks
  Other Names: sugar pill
  Arms: Sugar pill

SUMMARY:
The primary objectives of the study to evaluate the effects of two doses of nalbuphine HCl ER tablets on the change from baseline in the worst itch Numerical Rating Scale (NRS) in hemodialysis patients with moderate to severe uremic pruritus and to evaluate the safety and tolerability in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been receiving in-center hemodialysis for ≥ 3 months and are currently on a schedule of 3 times a week.
* Subject self-categorized themselves on the Patient Assessed Disease Severity Scale during Screening
* Subject meets standard of care hemodialysis efficiency guidelines during the three months prior to completing Screening
* Have demonstrated pruritus intensity on the Itch NRS during screening
* Male or female who are at least 18 years old at the time of Screening

Exclusion Criteria:

* Subject had a significant alteration in dialysis regimen during the Screening Period
* Subject receiving or anticipated to be receiving nocturnal dialysis or home hemodialysis treatment during the study.
* Subject has pruritus that is believed to be caused by a condition unrelated to end-stage renal disease
* Has had a history of substance abuse within 6 months prior to completing Screening
* Subject has a known drug allergy to opioids
* Subject is a pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (47):
- United States (41):
  - Nephrology Associates PC, Birmingham, Alabama
  - University South Alabama Medical Center, Mobile, Alabama
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - U.S. Renal Care Inc, Pine Bluff, Arkansas
  - North America Research Institute, Azusa, California
  - Pegasus Dialysis, LLC, Bakersfield, California
  - Central Nephrology Medical Group, Bakersfield, California
  - Academic Medical Research Institute, Los Angeles, California
  - Mark Lee MD, Inc, Whittier, California
  - Nephrology and Hypertension Associates PC, Middlebury, Connecticut
  - DaVita Inc Clinical Research Unit, Stamford, Connecticut
  - Nephrology Center DBA Paragon Health, Miami, Florida
  - Pines Clinical Research Inc, Pembroke Pines, Florida
  - Genesis Clinical Research, Tampa, Florida
  - DaVita Central Orlando Dialysis, Winter Park, Florida
  - Southwest Georgia Nephrology Clinic PC, Albany, Georgia
  - Renal Physicians of Georgia, Macon, Georgia
  - Pacific Renal Research Institute, Meridian, Idaho
  - Fresenius Medical Care of Evergreen Park, Evergreen Park, Illinois
  - Western New England Renal and Transplant Association, Springfield, Massachusetts
  - McComb Limited Care Facility, McComb, Mississippi
  - Kidney Associates of Kansas City PC, Kansas City, Missouri
  - Nephrology-Hypertension Associates of Central New Jersey PA, North Brunswick, New Jersey
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Newtown Dialysis Center, Inc, College Point, New York
  - DaVita Northtown's Dialysis Center, Tonawanda, New York
  - Durham Nephrology Associates, Durham, North Carolina
  - Wake Nephrology Associates PA, Raleigh, North Carolina
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - Nephrology Research Consortium, Bethlehem, Pennsylvania
  - Delaware Valley Nephrology, Philadelphia, Pennsylvania
  - Dialysis Clinic Inc., Philadelphia, Pennsylvania
  - South Carolina Nephrology and Hypertension, Hampton, South Carolina
  - South Carolina Nephrology and Hypertension, Orangeburg, South Carolina
  - Carolina Diabetes and Kidney Center, Sumter, South Carolina
  - Southwest Renal Research Institute, Chattanooga, Tennessee
  - U.S. Renal Care Inc, Fort Worth, Texas
  - U.S Renal Care Inc., Fort Worth, Texas
  - U.S. Renal Care Inc., Mansfield, Texas
  - Fresenius Medical Care Shorewood, Shorewood, Wisconsin
- Norbert Barlicki University Hospital No1. of the Medical University of Lodz, Lodz, Poland
- Romania (5):
  - International Healthcare Systems S.A IHS Craiova Dialysis Center, Craiova, Dolj
  - International Healthcare Systems S.A IHS Fundeni Dialysis Center, Bucharest
  - S.C Gral Medical S.R.L, Bucharest
  - S.C Diaverum Romania S.R.I, Industriilor Diaverum Dialysis Center, Bucharest
  - SC Diaverum Romania SRL, Splai Dialysis Center, Bucharest

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nalbuphine HCl ER 60mg | Nalbuphine HCl ER 120mg | Sugar Pill
Started | 128 | 120 | 125
Completed | 74 | 78 | 101
Not Completed | 54 | 42 | 24

BASELINE CHARACTERISTICS:
Population: Of the initial 373 participants randomized, 4 were never treated and, therefore, are not included in baseline demographic or frequency tables of treatment emrgent adverse events (TEAEs). Thus, the number of treated particpants was 369.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nalbuphine HCl ER 60mg | Nalbuphine HCl ER 120mg | Sugar Pill | Total
Number analyzed (Participants) | 126 | 120 | 123 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (12.1) | 55.2 (12.2) | 56.5 (13.0) | 55.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 51 | 49 | 158
  Male | 68 | 69 | 74 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 18 | 61
  Not Hispanic or Latino | 103 | 100 | 105 | 308
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3 | 6
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 66 | 55 | 60 | 181
  White | 57 | 62 | 59 | 178
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Europe | 23 | 23 | 23 | 69
  United States | 103 | 97 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Evaluation Period in Itch on the 0-10 Itch Numerical Rating Scale
Description: The evaluation period was defined as the average itch score over weeks 7 and 8 following initiation of treatment. A negative change form baseline (Evaluation Period - Baseline) signified inmprovement.
Time Frame: 8 weeks
Population: The sample sizes for each arm include participants who had a baseline value and at least one post baseline value for the average itch score during teh Evaluation Period.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nalbuphine HCl ER 60mg | Nalbuphine HCl ER 120mg | Sugar Pill
Number analyzed (Participants) | 82 | 84 | 108
units on a scale | -3.10 (2.35) | -3.49 (2.37) | -2.80 (2.22)

ADVERSE EVENTS:
Arm/Group | Nalbuphine HCl ER 60mg | Nalbuphine HCl ER 120mg | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/120 | 0/123
Serious Adverse Events (participants affected / at risk) | 16/126 | 8/120 | 19/123
Other Adverse Events (participants affected / at risk) | 0/126 | 0/120 | 0/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nalbuphine HCl ER 60mg (N=126) | Nalbuphine HCl ER 120mg (N=120) | Sugar Pill (N=123)
Cardiac failure congestive (Cardiac disorders) | 4 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Ilieus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Vertigo (Eye disorders) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No